CLINICAL TRIAL: NCT00503997
Title: Phase II Trial: Efficacy and Toxicity of Induction Pemetrexed (ALIMTA) and Oxaliplatin (ELOXATIN) in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Pemetrexed and Oxaliplatin in Treating Patients With Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jill Gilbert, MD, Associate Professor of Medicine; Director, Hematology/Oncology Fellowship Program; Section Chief, Solid Tumor Oncology; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC HN 0582; VU-VICC-HN-0582; VU-VICC-IRB-060100
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; untreated metastatic squamous neck cancer with occult primary
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Oxaliplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- drug therapy (Experimental)
  Interventions: Drug: oxaliplatin; Drug: pemetrexed disodium

INTERVENTIONS:
Drug: oxaliplatin — Group I: Patients receive pemetrexed disodium IV and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for up to 4 courses. If patient progresses before receiving 4 courses of treatment, treatment will be discontinued and patient will proceed to surgery.
  Group II: Patients receive treatment as in group I. If patient progresses before receiving 4 courses of treatment, treatment will be discontinued and patient will proceed to concurrent chemoradiotherapy.
  Other Names: Eloxatin
Drug: pemetrexed disodium — Group I: Patients receive pemetrexed disodium IV and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for up to 4 courses. If patient progresses before receiving 4 courses of treatment, treatment will be discontinued and patient will proceed to surgery.
  Group II: Patients receive treatment as in group I. If patient progresses before receiving 4 courses of treatment, treatment will be discontinued and patient will proceed to concurrent chemoradiotherapy.
  Other Names: Alimta

SUMMARY:
RATIONALE: Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving pemetrexed together with oxaliplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving pemetrexed together with oxaliplatin works in treating patients with locally advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the clinical response rate in patients with locally advanced squamous cell carcinoma of the head and neck treated with neoadjuvant pemetrexed disodium and oxaliplatin.

Secondary

* To evaluate the pathological complete response in patients who undergo surgical resection or post-induction biopsy.
* To assess toxicity of therapy, including the assessment of quality of life, fatigue, and head and neck cancer-related symptoms.
* To predict response and toxicities based on pharmacogenomics, genomics, and proteomics.

OUTLINE: This is a nonrandomized, open-label study. Patients are assigned to 1 of 2 groups based on resectability of disease (resectable vs nonresectable).

* Group I (resectable disease): Patients receive pemetrexed disodium IV and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for up to 4 courses. If patient progresses before receiving 4 courses of treatment, treatment will be discontinued and patient will proceed to surgery.

After completion of pemetrexed disodium and oxaliplatin, patients undergo surgical resection of disease.

* Group II (nonresectable disease): Patients receive treatment as in group I. If patient progresses before receiving 4 courses of treatment, treatment will be discontinued and patient will proceed to concurrent chemoradiotherapy.

After completion of pemetrexed disodium and oxaliplatin, patients undergo concurrent chemoradiotherapy.

Blood samples are collected at baseline and periodically during study for biomarker and pharmacokinetic studies.

Quality of life is assessed prior to each course of therapy and at 4-6 weeks after the last course.

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

Patients must meet all of the following criteria in order to be eligible for entry into the trial:

* Histologically or cytologically confirmed stage III - IVB HNSCC (includes unknown primary and ParaNasal Sinus cancers)but excludes nasopharyngeal, salivary gland or skin primaries (No TNM staging required)
* Patients must have a measurable disease defined by RECIST criteria
* Age > 18 years
* ECOG Performance Score of 0, 1 or 2
* Adequate bone marrow as evidenced by:

  * Absolute neutrophil count > 1,500/μL
  * Platelet count > 100,000/μL
* Adequate renal function as evidenced by serum creatinine < 1.5 mg/dL and CrCl > 45 mL/min as determined by calculated creatinine clearance using the Cockroft-Gault formula:

  * CrCl = (140-age) x (weight in kg)/72 x serum creatinine
  * Multiply by 0.85 (85%) for females
* Adequate hepatic function as evidenced by:

  * Serum total bilirubin < 1.5 mg/dL
  * Alkaline phosphatase < 3X the ULN for the reference lab
  * SGOT/SGPT < 3X the ULN for the reference lab
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial.
* Patients of childbearing potential and their partners must agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive, double barrier method or surgical intervention resulting in sterility).
* Patients must be able to interupt NSAIDs at 2 days before (5 days for long-acting NSAIDs),the day of, and 2 days following administration of Pemetrexed.
* Patients must be willing and able to take Folic Acid (350-1000 μg) daily beginning 1 week (7 days) prior to the first dose of Pemetrexed and continued daily until 3 weeks after the last dose of study therapy. In addition, patients must be willing to maintain a Pill Diary as part of study compliance.
* Patients must be willing and able to take Vitamin B12 (1000 μg) administered intramuscularly beginning 1 week (7 days) prior to the first dose of Pemetrexed and repeated at the planned End of Treatment visit (no later than 9 weeks from the first injection).
* Patients must be willing and able to take Dexamethasone (4 mg of oral or equivalent) that should be given twice daily on the day before, the day of, and the day after each dose of Pemetrexed for rash prophylaxis unless medically contraindicated.

Exclusion Criteria:

A patient may not be enrolled in the trial if any of the following criteria are met:

* Patients with an active infection or with a fever > 101.30 F within 3 days of the first scheduled day of protocol treatment
* History of prior malignancy within the past 3 years except for curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or localized prostate cancer with a current PSA of < 1.0 mg/dL on 2 successive evaluations, at least 3 months apart, with the most recent evaluation no more than 4 weeks prior to entry
* Patients with known hypersensitivity to any of the components of Oxaliplatin and Pemetrexed
* Patients who received any chemotherapy, radiation therapy or surgical resection other than diagnostic biopsies for HNSCC prior to the first scheduled day of protocol treatment
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment(investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Peripheral neuropathy ≥ Grade 2
* Patients who are pregnant or lactating
* Any other medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent,cooperate and participate in the study, or interferes with the interpretation of the results.
* History of allogeneic transplant
* Known HIV (active, previously treated or both)
* Presence of clinically detectable (by physical exam) third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage or other procedures prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Gilbert, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (7):
- United States (7):
  - Mitchell Memorial Cancer Center at Owensboro Medical Health System, Owensboro, Kentucky
  - Purchase Cancer Group - Paducah, Paducah, Kentucky
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Chung CH, Lee JW, Slebos RJ, Howard JD, Perez J, Kang H, Fertig EJ, Considine M, Gilbert J, Murphy BA, Nallur S, Paranjape T, Jordan RC, Garcia J, Burtness B, Forastiere AA, Weidhaas JB. A 3'-UTR KRAS-variant is associated with cisplatin resistance in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. Ann Oncol. 2014 Nov;25(11):2230-2236. doi: 10.1093/annonc/mdu367. Epub 2014 Jul 31. PMID 25081901
- [Derived] Psyrri A, Rampias T, Vermorken JB. The current and future impact of human papillomavirus on treatment of squamous cell carcinoma of the head and neck. Ann Oncol. 2014 Nov;25(11):2101-2115. doi: 10.1093/annonc/mdu265. Epub 2014 Jul 23. PMID 25057165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was open to accrual from 12/13/2006 to 4/9/2008.
Pre-assignment Details: This study consented 42 patients. One patient was found ineligible.
Groups:
- Pemetrexed/Oxaliplatin: Patients receive pemetrexed disodium IV and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for up to 4 courses. If patient progresses before receiving 4 courses of treatment, treatment will be discontinued and patient will proceed to surgery.
Period: Overall Study
Arm/Group | Pemetrexed/Oxaliplatin
Started | 42
Completed | 34
Not Completed | 8
Not completed — disease progression | 1
Not completed — Adverse Event | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed/Oxaliplatin
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Patient Response to Treatment Measured by RECIST Criteria
Description: RECIST response categories: Progressive disease (PD): >=20% increase in sum of longest diameter (LD) of target lesion(s), taking as reference smallest sum LD recorded since treatment started. Complete response (CR): disappearance of all target lesions. Partial response (PR): >=30% decrease in sum of LD of target lesion(s), taking as reference baseline sum LD. Stable disease (SD): neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD.
Time Frame: at 8 weeks
Measure: Number; unit: participants
Arm/Group | Pemetrexed/Oxaliplatin
Number analyzed (Participants) | 42
participants
  Complete Response | 1
  Partial Response | 18
  Stable Disease | 19
  Progressive Disease | 2
  Not Evaluable | 2

ADVERSE EVENTS:
Arm/Group | Pemetrexed/Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 7/42
Other Adverse Events (participants affected / at risk) | 11/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Oxaliplatin (N=42)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophagus pain (Gastrointestinal disorders) | 1 (1)
ANC/AGC (Investigations) | 1 (1)
hearing loss, sudden (Ear and labyrinth disorders) | 1 (1)
infection, port-a-cath (Infections and infestations) | 1 (1)
DVT/PE (Vascular disorders) | 1 (1)
myelosupression (Blood and lymphatic system disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
acidosis (Metabolism and nutrition disorders) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
malnutrition (Metabolism and nutrition disorders) | 1 (1)
obstructed PEG tube (Gastrointestinal disorders) | 1 (1)
tracheostomy tube changed (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cystitis (Renal and urinary disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
weight loss (Investigations) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Oxaliplatin (N=42)
hypokalemia (Metabolism and nutrition disorders) | 7 (7)
diarrhea (Gastrointestinal disorders) | 4 (4)
neutropenia (General disorders) | 7 (7)
dehydration (Gastrointestinal disorders) | 2 (2)
infection (Infections and infestations) | 2 (2)

LIMITATIONS AND CAVEATS:
The two cohorts of pemetrexed and oxaliplatin patients represented similar populations, thus the response data were combined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes